CLINICAL TRIAL: NCT05901519
Title: A Pilot Study of Liver Protection Using Prednisone for Patients Receiving Stereotactic Body Radiation Therapy for Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2022.120; HUM00234029 (Other: University of Michigan)
Record Dates: First submitted 2023-04-26; First posted 2023-06-13 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Radiation Therapy; Prednisone
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients treated with Prednisone (Experimental): Prednisone will be administered for three days before starting RT, and during the first three fractions of RT. Following an interim analysis of the decrease in sTNFR1 level, a decision will be made whether to administer prednisone for seven days prior to RT, and to continue for additional seven days during RT.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Patients will be treated with PO prednisone, once a day, at a dose of 60 mg/day

SUMMARY:
Patients on this study will self administer Prednisone for three days before starting Radiation Therapy (RT) and continue to take 60 mg/day during the first three fractions of RT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatocellular carcinoma are eligible for this trial. Hepatocellular carcinoma is defined as having at least one of the following:

  1. Biopsy proven hepatocellular carcinoma (HCC); or
  2. A discrete hepatic tumor(s) as defined by the AASLD criteria (80) - for cirrhotic patients, >1cm with arterial hypervascularity and venous or delayed phase washout on contrast enhanced CT or MRI.
* Patients must have recovered from the acute effects of prior liver-directed therapy (e.g., RT, RFA, or TACE), and a minimum of 4 weeks must have passed since the last procedure and protocol therapy.
* Patients must have a performance status of ≤2.
* Patients must be 18 years of age or older.
* Patients with at least one of the following:

  1. ALBI score equal to (-1.81) or higher (worse). This value was calculated as the equivalent ALBI score for CP score equal 7 in Cousins et al study's cohort(59).
  2. Lesion(s) with a cumulative treatment diameter of ≥ 4cm.
  3. CP score equal to 7 or higher (worse).
* Patients must understand and be willing to sign an informed consent form approved for this purpose by the Institutional Review Board (IRB) of the University of Michigan Medical Center indicating that they are aware of the investigational aspects of the treatment and the potential risks.

Exclusion Criteria:

* Any serious disease, comorbidity or intercurrent illness which precludes delivery of radiation therapy, as determined by the treating investigator.
* Any contraindication to the administration of steroids, including

  * Documented hypersensitivity to prednisone or any component of the formulation.
  * Systemic fungal infection.
  * Patients with uncontrolled infections or with chronic infections requiring antibiotics.

Infections are considered controlled if appropriate therapy has been instituted and, at the time of enrollment, no signs of progression are present. Progression of infection is defined as hemodynamic instability attributable to sepsis, new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.

* Uncontrolled hyperglycemia.

  * Patients with insulin -dependent diabetes.
  * Patients with decompensated liver disease, defined as: clinical ascites requiring paracentesis, hepatic encephalopathy, hepatorenal syndrome or variceal hemorrhage.
  * Active gastrointestinal bleeding within 30 days of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mitigation of liver inflammation as reflected by sTNFR1 levels | at baseline, day of first RT fraction, day of 3rd RT fraction and at 1-, 3- and 6-months post commencing radiation therapy
  Measuring whether sTNFR1 level is attenuated following prednisone treatment, given before and during radiation therapy for HCC patients who are at high risk of radiation induced liver toxicity. sTNFR1 levels will be summarized descriptively at each time point as absolute values and change from baseline (prior to taking prednisone). Longitudinal regression models will be used to test whether mean changes over time are statistically significant. Treatment with prednisone will be considered successful if it causes a decrease in the level of sTNFR1 of 50%, which would be predicted to decrease toxicity by 15%.

SECONDARY OUTCOMES:
Estimating the safety of the steroid treatment | up to 6 weeks from start of study treatment
  Define steroid administration protocol based on the rate of drug-related grade 3-5 adverse events attributable to the study drug and experienced within the first 6 weeks of study treatment. These will be assessed via NCI's CTCAE version 5.0. Toxicity rates for patients on this study will be compared to a propensity matched historical control cohort of recently treated patients at UM who were not treated with prednisone.
Percent of patients who complete of the proposed steroid treatment | up to 6 weeks from start of study treatment
  Successful completion of steroid treatment.
Evaluate whether steroid treatment reduces radiation-induced liver toxicity | up to 6 weeks from start of study treatment
  Rate of liver decompensation (as measured by worsening in ALBI score>0.5) or grade 3-5 GI bleeding during the subsequent 6 months following radiation treatment. The former are laboratory values that are already collected as part of standard of care. The latter will be assessed via the NCI CTCAE version 5.
Assess whether steroids have a durable ability to attenuate the level of inflammation as reflected by sTNFR1 level | up to 6 months from start of study treatment
  Determining the mitigation of the inflammatory state, as reflected by biomarkers previously proposed in the literature to correlate with radiation-induced liver injury.
Assess tumor response | up to 6 months from start of study treatment
  assessing tumor response as part of standard of care to determine response rate

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Lawrence, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- Rogel Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No